CLINICAL TRIAL: NCT01909648
Title: HbA2 Leuven and Its Impact on HbA1c Results
Acronym: HbA2 Leuven
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S55709; S55709 (Other: UZLeuven)
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Family Study HbA2 Leuven Mutation.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HbA2 Leuven (Other): Presence of HbA2 Leuven mutation, demonstrated by molecular diagnosis on blood sample.
  Interventions: Other: Blood withdrawal; Genetic: Blood withdrawal

INTERVENTIONS:
Other: Blood withdrawal
  Other Names: Impact of mutation on routine HbA1c measurements.
Genetic: Blood withdrawal
  Other Names: Demonstration of HbA2 Leuven mutation

SUMMARY:
The study is designed to demonstrate HbA2 Leuven mutation and to asssess its impact on routine HbA1c measurements.

DETAILED DESCRIPTION:
HbA2 Leuven mutation will be investigated using molecular diagnostic techniques.

Interference on HbA1c measurements will be assessed in HbA2 Leuven carriers using different methodologies.

ELIGIBILITY:
Inclusion Criteria:

* Family history of HbA2 Leuven mutation.

Exclusion Criteria:

* Any condition inhibiting simple blood withdrawal.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Demonstration of presence/absence of HbA2 Leuven mutation | 1 year

SECONDARY OUTCOMES:
Demonstration of impact of HbA2 Leuven mutation on routine HbA1c measurements | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Davy MJ Kieffer, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Pieter Gillard, MD, PhD, Study Chair — Universitaire Ziekenhuizen KU Leuven; Koen Desmet, PharmD, Study Chair — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium